CLINICAL TRIAL: NCT03526588
Title: Umbilical Cord Blood Mononuclear Cells for Hypoxic Neurologic Injury in Infants With Congenital Diaphragmatic Hernia (CDH)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Competing randomized trial of an experimental therapy limited initial enrollment. The trial was completed, published, and the experimental therapy became broadly desired. Given this, the investigators felt it best to terminate this competing study.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Medical Center Regenerative Medicine Consortium (Unknown)
Responsible Party: Principal Investigator, Matthew T Harting, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0148
Record Dates: First submitted 2018-04-27; First posted 2018-05-16 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: CDH
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous umbilical cord blood (Experimental)
  Interventions: Biological: Autologous umbilical cord blood

INTERVENTIONS:
Biological: Autologous umbilical cord blood — 6×10^6 mononuclear cells isolated from the patient's own umbilical cord blood per dose. 4 total doses administered intravenously over 7 days.

SUMMARY:
The purpose of this study is to investigate the use of autologous umbilical cord blood (UCB) mononuclear cells to mitigate hypoxic neurologic injury among infants with high-risk congenital diaphragmatic hernia (CDH).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CDH between 20 and 36 weeks estimated gestational age (EGA)
* Only one of the following fetal criteria and one of the following postnatal criteria must be met for enrollment. Fetal criteria: an ultrasound (US)-obtained observed to expected lung to head ratio (o/e LHR) less than or equal to 35% or 2) a fetal magnetic resonance imaging (fMRI)- obtained observed to expected total fetal lung volume (o/e TFLV) less than or equal to 35%. Postnatal criteria: 1) Cord blood gas (CBG) with potenital hydrogen (pH) <7.0, 2) Arterial blood gas (ABG) with pH <7.2 on 2 gasses within the first 24 hours, 3) Preductal oxygen saturation (O2 sat) <90% x 2 total hours (not necessarily consecutive) within the first 24 hours, or 4) Oxygenation Index (OI) >20 x 2 total hours (not necessarily consecutive) within the first 24 hours.

Exclusion Criteria:

* Genetic/chromosomal abnormality: Trisomy 21, Trisomy 18, Trisomy 13 or other, significant genetic abnormality. Microdeletions or other mild genetic abnormalities are not considered exclusionary.
* Severe/major cardiac anomaly: coarctation of the aorta, combined atrial and ventricular septal defects, hypoplastic left heart syndrome, tetralogy of fallot, double outlet right ventricle, atrioventricular canal defects, or other hemodynamically significant defects.
* Moderate/severe neurologic / intracranial abnormality: Grade III or IV intraparenchymal hemorrhage, space occupying mass or lesion, or clinically significant traumatic lesion such as a subdural or epidural hemorrhage.
* Prematurity <30 weeks estimated gestational age (EGA): Birth at 29 6/7 weeks or before
* Participation in an alternative prenatal intervention study: Fetoscopic Endotracheal Occlusion (FETO)
* Unwillingness / inability to return for follow-up evaluation and assessment

Ages: 10 Minutes to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by vital sign monitoring (heart rate) | daily for 7 days following the initial infusion
Safety as assessed by vital sign monitoring (systolic blood pressure) | daily for 7 days following the initial infusion
Safety as assessed by vital sign monitoring (diastolic blood pressure) | daily for 7 days following the initial infusion
Safety as assessed by vital sign monitoring (temperature) | daily for 7 days following the initial infusion
Safety as assessed by pulmonary status (indicated by peak inspiratory pressure (PIP)) | daily for 7 days following the initial infusion
Safety as assessed by pulmonary status (indicated by positive end expiratory pressure (PEEP)) | daily for 7 days following the initial infusion
Safety as assessed by pulmonary status (indicated by respiratory rate (RR)) | daily for 7 days following the initial infusion
Safety as assessed by pulmonary status (indicated by Fraction of inspired oxygen (FiO2)) | daily for 7 days following the initial infusion
Safety as assessed by presence of new infiltrates or altered aeration upon chest radiography | daily for 7 days following the initial infusion
Safety as assessed by cardiovascular status (indicated by heart rate) | daily for 7 days following the initial infusion
Safety as assessed by cardiovascular status (indicated by systolic blood pressure) | daily for 7 days following the initial infusion
Safety as assessed by cardiovascular status (indicated by diastolic blood pressure) | daily for 7 days following the initial infusion
Safety as assessed by cardiovascular status (indicated by changes in cardiovascular pharmacologic support) | daily for 7 days following the initial infusion
Safety as assessed by infection status (indicated by body temperature) | daily for 7 days following the initial infusion
Safety as assessed by infection status (indicated by white blood cell count) | 7 days following the initial infusion
Safety as assessed by infection status (indicated by physical signs of infection) | daily for 7 days following the initial infusion
Safety as assessed by liver function (indicated by Alanine aminotransferase (ALT) levels) | 7 days following the initial infusion
Safety as assessed by liver function (indicated by aspartate aminotransferase (AST) levels | 7 days following the initial infusion
Safety as assessed by liver function (indicated by bilirubin levels) | 7 days following the initial infusion
Safety as assessed by liver function (indicated by albumin levels) | 7 days following the initial infusion
Safety as assessed by blood urea nitrogen (BUN) levels | 7 days following the initial infusion
Safety as assessed by creatinine levels | 7 days following the initial infusion
Safety as assessed by carbon dioxide (CO2) levels | 7 days following the initial infusion
Safety as assessed by glucose levels | 7 days following the initial infusion
Safety as assessed by serum chloride levels | 7 days following the initial infusion
Safety as assessed by serum potassium levels | 7 days following the initial infusion
Safety as assessed by serum sodium levels | 7 days following the initial infusion
Neurologic/neurodevelopmental status as assessed by intracranial abnormalities upon magnetic resonance imaging (MRI) | within 14 days of discharge (discharge occurs at about 2-4 months after birth)
Neurologic/neurodevelopmental status as assessed by receipt of neurologic pharmacologic medications | at the time of discharge (which is about 2-4 months after birth)
Neurologic/neurodevelopmental status as assessed by Bayley Scales of Infant and Toddler Development-III (BSID-III) | 2 years after birth
  The Bayley-III is an individually-administered examination that assesses the current developmental functioning of infants and young children from birth to 42 months of age. The Bayley is a standardized, norm-referenced measure that assesses development in Cognitive, Language and Motor domains. Composite standard scores can be derived that have a mean of 100 and a standard deviation of 15.

SECONDARY OUTCOMES:
Mortality | 2 years after birth
Length of stay in hospital | from birth to discharge or death, whichever occurs first (discharge occurs at about 2-4 months after birth)
Progression of pulmonary hypertension as assessed by echocardiography | within 24 hours of birth, prior to operative repair (occurs between day 2 & 14 of life), prior to discharge (usually 2-6 months), and after discharge (2wks-6 months following discharge)
Duration of extracorporeal membrane oxygenation (ECMO) support | days from ECMO initiation until decannulation (an average of 3 weeks)
Duration of ventilatory support | from initiation of ventilation until extubation (an average of 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T. Harting, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- See also: The Comprehensive Center for CDH Care at Children's Memorial Hermann Hospital and The University of Texas Health Science Center in Houston (Texas Medical Center) — http://childrens.memorialhermann.org/conditions/cdh-treatment/